CLINICAL TRIAL: NCT03119974
Title: Rate of Prolonged Response After Stopping Thrombopoietin-receptor Agonists Treatment in Immune Thrombocytopenia: a Prospective Multicenter Open Study
Brief Title: Rate of Prolonged Response After Stopping Thrombopoietin-receptor Agonists Treatment in ITP
Acronym: STOP-AGO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P150956; 2016-001786-93 (EudraCT Number)
Record Dates: First submitted 2016-12-23; First posted 2017-04-19 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Persistent or Chronic ITP
Keywords: ITP; TPO-RAS; Thrombopoietin-receptor agonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tpo-RA discontinuation (Other)
  Interventions: Drug: Tpo-RA discontinuation

INTERVENTIONS:
Drug: Tpo-RA discontinuation — a standardized strategy of dosage reduction will be implemented according to a predetermined scheme on persistent and/or chronic ITP patients who have previously achieved a stable and prolonged (> 2 months) complete response (platelets counts > 100 x 109/L) period on Tpo-RA treatment.

SUMMARY:
Thrombopoietin-receptor agonists (Tpo-RAs) have profoundly changed the management of ITP. However, today, there are no international recommendations concerning the long-term use of these costly, potentially pro-thrombotic agents, and that could induce bone marrow fibrosis in case of prolonged treatment. Tpo-RAs have been thought to play only a supporting role in ITP management. But our center along with many other research centers, have reported unexpected cases of durable remission after Tpo-RAs discontinuation in adult chronic ITP. In these retrospective studies, more than 20 % of patients were able to achieve prolonged remission.

The purpose of this study is to demonstrate that a substantial proportion of ITP patients may achieve a prolonged response after Tpo-RA discontinuation.

The investigators developed, in this study, a standardized procedure to discontinue Eltrombopag and Romiplostim, wherein the dose will be slowly tapered to limit the risk of bleeding. In case of relapse after Tpo-RA discontinuation, the decision to start a new therapy will be based on the clinician's judgment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Diagnosis of ITP according to the standard definition
3. Disease duration of more than 3 months at Tpo-RA initiation
4. Platelet count > 100 x 109/L for more than 2 months on Tpo-RA Therapy, with at least 3 platelet counts > 100 x 109/L
5. Blood count lasting for less than 7 days
6. Normal marrow aspirate for patients aged of 60 and over
7. Informed signed consent
8. Treatment with Tpo-RA for at least 3 months

Exclusion Criteria:

1) Anticoagulation or anti-platelet treatment 2) Recent treatment with corticosteroids ± intravenous immunoglobulins (less than 2 months) 3) Rituximab or splenectomy within the 2 months preceding the Tpo-RA initiation 4) Rituximab or splenectomy after Tpo-RA initiation/RA initiation 5) Previous failure of Tpo-RA discontinuation 6) Pregnant or breastfeeding women 7) No affiliation to a social security scheme or other social protection scheme 8) Inability or refusal to understand or refusal to sign the informed consent from study participation 9) Patient deprived of freedom or under legal protection (guardianship, curatorship) 10) Hypersensitivity to Romiplostin or to any of the excipients or to E. coli derived proteins

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieving an overall response (complete response and response) at week 24 (6 months). The criteria of response will be defined according to international terminology | week 24 (6 months)
  the criteria of response will be defined as the following:
  * Response (R) will be defined as sustained platelet count >30x109/L in the absence of bleeding or use of any other ITP directed therapies between the week 0 (discontinuation) and week 24.
  * Complete response (CR) by a platelet count > 100x 109/L in the absence use of any other ITP directed therapies between week 0 and week 24.
  * Patients will be considered as being non-responders (NR) if:
    1. Their platelet count is < 30 x 109/L between week 0 and week 24, but also, in the setting of this study if:
    2. They need a rescue therapy (a new course of corticosteroids and/or intravenous immunoglobulin) after inclusion.

SECONDARY OUTCOMES:
The rate of overall response after Tpo-RAs discontinuation | 24 and 52 weeks
  response and complete response
The duration of overall response after Tpo-RAs discontinuation. | 24 and 52 weeks
  response and complete response
The number of bleeding events during the reduction period and along the study period at weeks 4, 8, 12,24,36, 52 | at weeks 4, 8, 12,24,36, 52
  Safety assess of Tpo-RAs discontinuation
The rate of the response to a new course of Tpo-RAs in case of relapse after Tpo-RAs discontinuation at one year | 52 weeks
  Rate of the response in case of relapse
The delay of the response to a new course of Tpo-RAs in case of relapse after Tpo-RAs discontinuation | 52 weeks
  Delay of the response in case of relapse
To identify predictive factors, for overall prolonged response | Weeks 24
  Search for predictive factor of response

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Mahevas, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri-Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cottu A, Guillet S, Viallard JF, Riviere E, Cheze S, Gobert D, Neel A, Graveleau J, Marolleau JP, Lefrere F, Moulis G, Lega JC, Moignet-Autrel A, Robbins A, Crickx E, Boutin E, Noel N, Malphettes M, Galicier L, Audia S, Bonnotte B, Lambotte O, Fain O, Gerfaud-Valentin M, Terriou L, Martis N, Morin AS, Perlat A, Le Gallou T, Roy-Peaud F, Puyade M, Comont T, Limal N, Languille L, Michel M, Godeau B, Mahevas M. Long-term follow-up of the STOPAGO study. Blood. 2025 Jan 9;145(2):244-247. doi: 10.1182/blood.2024025707. PMID 39476101
- [Derived] Guillet S, Crickx E, Azzaoui I, Chappert P, Boutin E, Viallard JF, Riviere E, Gobert D, Galicier L, Malphettes M, Cheze S, Lefrere F, Audia S, Bonnotte B, Lambotte O, Noel N, Fain O, Moulis G, Hamidou M, Gerfaud-Valentin M, Marolleau JP, Terriou L, Martis N, Morin AS, Perlat A, Le Gallou T, Roy-Peaud F, Robbins A, Lega JC, Puyade M, Comont T, Limal N, Languille L, Zarrour A, Luka M, Menager M, Belmondo T, Hue S, Canoui-Poitrine F, Michel M, Godeau B, Mahevas M. Prolonged response after TPO-RA discontinuation in primary ITP: results of a prospective multicenter study. Blood. 2023 Jun 8;141(23):2867-2877. doi: 10.1182/blood.2022018665. PMID 36893453